CLINICAL TRIAL: NCT04817735
Title: Calcium Algorithm Sizing for bicusPid Aortic Valve Evaluation With Raphe: the CASPER Registry
Brief Title: The CASPER Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Sonia Petronio, Professor, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI-2021-01
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Bicuspid Aortic Valve
Keywords: TAVI; MSCT; Bicuspid
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other)
  Interventions: Procedure: TAVI

INTERVENTIONS:
Procedure: TAVI — TAVI sizing with dedicated algorithm

SUMMARY:
The CASPER study is a prospective, international, multicenter registry which aims to evaluate the use of an algorithm for choosing the size of the prosthesis to be implanted in patients with bicuspid aortic stenosis type I treated by TAVI with Evolut® Pro prostheses (23 -26-29) and Evolut® R 34.

DETAILED DESCRIPTION:
STUDY DESIGN

This is an Investigator initiated, international, multicenter, prospective registry, enrolling 100 consecutive BAV patients who will undergo TAVI with the Evolut R/Pro (23-26-29)/Evolut R 34THV.

Enrollment will be without limitation for each center (competitive enrollment). The indication for TAVI will be based on each local Heart Team decision. As per local institution's regulatory policy, each patient will provide a written informed consent for the TAVI procedure, anonymous data collection and analysis. Each center will use its own consent template.

All data will be collected in an electronic clinical report form (eCRF).

STUDY POPULATION Population

All consecutive patients diagnosed with type 0 or type 1 bicuspid aortic valve stenosis or steno-insufficiency disease, undergoing transcatheter aortic valve implantation, as per local standard of care.

CASPER algorithm

The sizing of the THV will be performed according to the proposed algorithm.

First step ("calcium impact"): subtract 1 mm in patients with aortic calcium volume ≥300 mm3 (i.e. ≥ Class I); no subtraction in patients with aortic calcium volume <300 mm3 (i.e. Class 0).

Second step ("raphe impact"): subtract 1 mm if the raphe length is ≥50% of the perimeter derived mean annulus diameter Further 0.5 mm will be subtracted if a high burden of calcium is distributed predominantly on the raphe site.

In case of bicuspid Type 0 the second step should be skipped.

Transcatheter Aortic Valve Implantation Procedure

TAVI will be performed according to the local standards of care. Balloon valvuloplastywill be performed to prepare for TAVI deployment, at operator's discretion. Balloon size should not exceed the minimal diameter of the aortic annulus at baseline.

TAVI deployment will be performed as the current best practices. All Centers will be encouraged to implant THV according to the two cusp alignment technique. If necessary, post dilatation will be performed, based on the final hemodynamics and aortic regurgitation assessment. The postdilatation will be performed according to the calcium burden with a balloon size diameter equal to the minor annulus diameter or to the mean diameter.

Post-procedural MSCT scan

The post-procedural MSCT scan must be performed between 2 and 30 days after the index procedure.

Post implant measurements of THV dimensions (perimeter and area) will be obtained at inflow level, raphe level, and stent waist level (defined as the smallest dimension observed at any plane of the implanted prosthesis). If the raphe level corresponds to the stent waist level, only one measurement will be reported.

Eccentricity index will be calculated for each level. Eccentricity will be defined as 1-(minimal diameter/maximal diameter) and will be calculated both at the inflow and at the narrowest level.

The post-procedural raphe length (defined as the longest measurable dimension of the structure) will be measured at the same level of pre-procedural MSCT. The ratio between the pre and post-procedure raphe length will be calculated for the assessment of raphe shortening.

Strut separation data will be acquired (maximal strut distance, mean strut distance, strut eccentricity index, i.e. maximal-minimal strut separation). The stent strut spaces will be measured separately at the inflow level, with the first stent strut defined as the strut closest to the commissure between the non-coronary and right coronary sinuses. The subsequent struts will be numbered clockwise in an ascending order (1-15 for the Evolut THV).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. NYHA≥2 and/or syncope and/or angina.
3. Patient judged by the Heart Team as indicated for TAVI.
4. Anatomical suitability for transfemoral or any alternative access TAVI, based on MSCT assessment and local expertise and preference.
5. Estimated life expectancy>1 year.

Exclusion Criteria:

1. Age <18 years
2. Estimated life expectancy<1 year
3. Pure aortic regurgitation.
4. LVEF<20%
5. No baseline MSCT evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of the CASPER algorithm | 1 year
  The objective of the study is to validate the CASPER algorithm in a prospective cohort using a self-expandable THV, in order to assess the safety and efficacy of bicuspid aortic valve sizing based on calcium burden and raphe length.

SECONDARY OUTCOMES:
Safety of the CASPER algorithm | 1 year
  To assess valve performance in terms of prosthesis mismatch and valve dysfunction (clinical features), and post-procedural CT assessment of the prosthesis behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No